CLINICAL TRIAL: NCT04878445
Title: A Tissue Engineering Approach to Improve Lung Function and Clinical Outcome in Patients With COPD
Brief Title: Tissue Engineering Approaches to Treat COPD
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1517
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung cells, including DASCp63/Krt5 with a possible role in disease pathology, will be isolated, expanded in vitro, characterised, and banked. Biomaterials will be selected and tested with regards to mechanical and physical properties and selected for use in the production of TELEs with properties matched to healthy and diseased lung tissue.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: 10 participants with no COPD: Control patients Have no physician diagnosis of COPD Have no other significant chronic lung disease (asthma, fibrotic diseases) or ongoing lung infection other than the suspected cancer for which they have been referred for surgery.
  Lifelong never-smokers or ex-smokers (< 10 pack years). (1 pack year= 20 cigarettes/day for 1 year).
  Interventions: Procedure: Patients undergoing standard surgery, excess tissue only will be analysed with patient consent.
- Cohort B: 10 participants with COPD - chronic bronchitis: Have a physician diagnosis of COPD with primarily a chronic bronchitis presentation (determined via CT, spirometry, histopathology, GOLD COPD classification).
  Interventions: Procedure: Patients undergoing standard surgery, excess tissue only will be analysed with patient consent.
- Cohort C: 10 participants with COPD emphysema: Have a physician diagnosis of COPD with primarily a emphysema presentation (determined via CT, spirometry, histopathology, GOLD COPD classification) .
  Interventions: Procedure: Patients undergoing standard surgery, excess tissue only will be analysed with patient consent.

INTERVENTIONS:
Procedure: Patients undergoing standard surgery, excess tissue only will be analysed with patient consent. — Lung samples will be obtained from surplus, healthy margin lung tissue resected from patients with suspected or confirmed lung cancer or from resected tissue from lung volume reduction surgery.

SUMMARY:
The study is a pilot/laboratory study comparing lung tissue from control participants with tissue from COPD participants with a chronic bronchitis or emphysema phenotypes. Tissue will be characterised mechanically and biochemically.

Lung cells, including DASCp63/Krt5 with a possible role in disease pathology, will be isolated, expanded in vitro, characterised, and banked. Biomaterials will be selected and tested with regards to mechanical and physical properties and selected for use in the production of TELEs with properties matched to healthy and diseased lung tissue.

The resulting TELEs will be tested in an ex vivo tissue culture model to determine the extent of their integration with lung.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is currently ranked as the third leading cause of death with an annual associated global healthcare cost of £1.3 trillion (1). It is the second most common cause of emergency hospital admissions with high morbidity and mortality. COPD results in a progressive loss of lung function, leading to respiratory failure. This loss of lung function is associated with repetitive cycles of inflammation and parenchymal scarring leading to the development of emphysema. This is a consequence of the breakdown of the delicate parenchymal structures and lung remodelling, with accumulation of fibrous tissue and loss of the alveolar-capillary functional units that are essential for effective gas exchange. Macroscopically the lungs become stiffer and unable to support the patient through the physiological inhalation/exhalation breathing cycles (2).

The presence of emphysema also results in the loss of lung elastic recoil as pockets of air form in place of damaged bronchioles and alveoli reducing the available volume for the next inhalation. The collapse of the airways during exhalation leads to increased lung volumes causing hyperinflation and gas trapping. Patients become progressively symptomatic with increasing breathlessness, reduced exercise tolerance and poor quality of life.

The pharmacological treatment options for emphysema are limited; current therapy aims to improve airflow limitation, reduce airway inflammation and reduce exacerbations, but does not reverse lung damage (3). Lung transplantation and lung volume reduction surgery (LVRS) is available for a selected minority of patients with severe emphysema. The recent introduction of non-invasive endoscopic mechanical treatment with Valves reduces severely damaged lung volume and re-directs air to the healthier tissue while Coils improves elastic lung recoil (4, 5). These interventions however do not improve survival.

Previous work performed within our laboratories has determined that hydrogel/elastin-based constructs can achieve mechanical values consistent with those of the alveolar wall when seeded with lung fibroblasts (1). This raises the intriguing question of whether tissue-engineered constructs (TEC) could be used to restore mechanical integrity of the emphysematous lung, via air pocket displacement and local integration, and ultimately by regeneration of local lung architecture.

Coupled to the work described above a recent observation went some way to detailing the mechanism behind the previously misunderstood, but physiologically critical, capacity for lung tissue to regenerate following on from acute disease such as pneumonia or acute respiratory distress syndrome (6). The key appears to lie with a population of distal airway stem cells who co-express Trp63 (p63) and Keratin 5 (Krt5). These DASCp63/Krt5 cells appear to migrate to sites of injury in the lung where they have demonstrated differentiation capacity including lineages such as type I and II pneumocytes and bronchiolar secretory cells. It is crucial to our understanding of chronic lung disorders, and design of future cell-based therapies, whether these cells remain present and dormant in diseased lung tissue or lost through as yet unknown mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged over 18 years- .
* Must be competent to give written informed consent.
* Scheduled to undergo clinical indicated surgery to remove lung tissue.

Exclusion Criteria:

* Patient unable to give informed consent
* Significant long term condition or lung pathology (infection, asthma, fibrotic lung diseases) other than that for which they have been referred for surgery.

Post Surgery

• Insufficient tissue removed to supply the laboratory study after consultation with the Consultant histopathologist.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic obstructive pulmonary disease (COPD) is currently ranked as the third leading cause of death with an annual associated global healthcare cost of £1.3 trillion. It is the second most common cause of emergency hospital admissions with high morbidity and mortality. COPD results in a progressive loss of lung function, leading to respiratory failure. This loss of lung function is associated with repetitive cycles of inflammation and parenchymal scarring leading to the development of emphysema. This is a consequence of the breakdown of the delicate parenchymal structures and lung remodelling, with accumulation of fibrous tissue and loss of the alveolar-capillary functional units that are essential for effective gas exchange. Macroscopically the lungs become stiffer and unable to support the patient through the physiological inhalation/exhalation breathing cycles.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-08-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The overall aim of this project is to produce in vitro tissue engineered lung equivalents (TELEs) seeded with cells obtained from: | Through study completion upto 1 year
  P1) The determination of the scale-up suitability of in vitro lung equivalents, their mechanical properties, and in vitro degradation rates.
  P2) Development of in vitro DASCp63/Krt5 culture models to support re-establishment of local lung architecture.
  P3) Establishment of ex vivo lung culture models to support the lung tissue equivalents' evaluation.

SECONDARY OUTCOMES:
To achieve an understanding of the mechanical properties of diseased and healthy lung tissue. | Through study completion, upto 1 year
  To evaluate and tune hydrogel or foamed biomaterials to identify compositions which reflect the properties of healthy and diseased lung tissue.
  S3) Creation of lung cell banks e.g. fibroblasts, pneumocytes, club cells, from diseased and healthy tissue.
  S4). The identification of the presence/absence of DASCp63/Krt5 in healthy/diseased lung tissue and disease-association with retention of properties.
  S5). Insertion of tissue engineered lung pieces into ex vivo lung slice culture and evaluation of cell spreading and construct integration.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, Staffordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No